CLINICAL TRIAL: NCT06779838
Title: Randomised Controlled Trial (RCT) to Assess the Feasibility, Acceptability and Preliminary Effectiveness of Group Emotion-focused Therapy (EFT) Intervention for Transdiagnostic Eating Disorders/Difficulties in Student Counselling Services.
Brief Title: Effectiveness of Group EFT for Transdiagnostic Eating Disorders/Difficulties Within Student Counselling Services.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETH2324-0310
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa; Bulimia; Binge Eating Disorder; Eating Disorder Not Otherwise Specified; Eating Disorder Symptom and Body Image Dissatisfaction
Keywords: Emotion focused therapy; eating disorder; body weight shape concerns; university counselling services; group emotion focused therapy; inner critic eating disorder; transdiagnostic eating disorders
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the intervention group or a treatment as usual control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: group emotion focused therapy intervention (Experimental): The intervention is a 10 to 12-week (depending on number of participants recruited [intervention is n+2 weeks long] closed therapy group for students seeking support regarding issues related to eating, weight and shape concerns. Group members will be facilitated to recognise and explore some of the difficult emotions underlying these issues. In particular, the group will focus on 'taming' the inner critic, that part of ourselves that criticises or chastises us for not being good enough. By identifying the critic in ourselves and by witnessing it in others, group members may be better positioned to figure out what they really need from themselves at times of difficulty. There will be some information provided around eating and emotions, with the focus of the sessions being on experiential exercises under the guidance of the group facilitators.
  Interventions: Other: Group Emotion Focused Therapy Intervention
- Control: treatment as usual (Active Comparator): Students assigned to this arm will engage with the university counselling service as usual. This could include individual counselling, attending groups within the service or signposting to external agencies. Participants will be asked to state what support they have accessed.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: Group Emotion Focused Therapy Intervention — The EFT group intervention: Taming the Inner Critic: Emotion-Focused Group Therapy for Eating and Body Concerns. This group is a 10-12 week (number of participants=8-10 +2 sessions) closed therapy group for students seeking support regarding issues related to eating and/or body concerns. Working one-to-one and within the group, group members will be facilitated to recognise and explore some of the difficult emotions underlying and driving eating and/or body related issues. In particular, the group will focus on 'taming' the inner critic, that part of ourselves that criticises or chastises us for not being good enough. By identifying the critic in ourselves and by witnessing it in others, group members will be better positioned to figure out what they really need from themselves at times of difficulty, and thus better able to access self-compassion and self-assertion. There will be some psychoeducation, both around eating and emotions, but this will be largely in a handout format, with
  Arms: Treatment: group emotion focused therapy intervention
Other: Treatment as Usual (TAU) — Treatment that would otherwise be offered by the university counselling service (one on one counselling, a group, or signposting to external support).
  Arms: Control: treatment as usual

SUMMARY:
What is the purpose of the study? Emotion-Focused Therapy (EFT) is a therapeutic approach that helps individuals identify, explore, and transform difficult emotions to improve emotional wellbeing and resolve psychological issues. While there is a growing body of evidence for the effectiveness of both individual and group EFT with a range of difficulties, including eating disorders, this has not yet been sufficiently explored within university counselling services. The purpose of this study is to assess the feasibility, acceptability, and preliminary effectiveness of a group EFT intervention for students experiencing eating disorders or concerns related to eating, weight, and shape. The study aims to determine whether this type of therapy can be effectively delivered within a university counselling service, and if it could potentially improve participants' mental health and wellbeing.

DETAILED DESCRIPTION:
Who is being asked to participate? You are invited to participate if you: are experiencing an eating disorder or have eating, weight and shape concerns, have a body mass index greater than 15kg/m2 and have sufficient English for talking therapy. You will be ineligible to take part if you: are participating in psychological one-to-one or group therapy at the same time as attending the intervention group, have considerable psychological risk, including active suicidal plans, are experiencing psychosis, have an alcohol or substance use issue, pose a risk of harm towards others, are pregnant, or have a diagnosed intellectual disability that impairs your ability to access therapy.

Do I have to take part? Your participation in this study is entirely voluntary. If you agree to take part, I will then ask you to complete a consent form. You are free to withdraw at any time, without giving a reason.

Randomised Controlled Trial (RCT) The study will use an RCT design, meaning that, if you sign up for the study, you will be randomly assigned either to partake in the group EFT intervention, or to not partake in this. Regardless of the group to which you are assigned, you will be asked to complete sets of questionnaires at the beginning and end of the study. This will allow us to compare questionnaire data for those who received the intervention and those who did not, to gain an initial indication of whether the intervention is helpful or not. Your engagement is therefore of significant value to us regardless of whether you take part in the intervention during the study period.

What will happen to me if I take part? You will first undergo a screening process to ensure that you meet the eligibility criteria. If you are eligible, you will be randomly assigned to either the intervention group, which will participate in the EFT group therapy, or to the control group, who will not participate in the EFT group therapy. . There is an equal chance of being put into either group. Both groups will be asked to complete a set of questionnaires before and after the intervention period, regardless of group assignment. The questionnaires will measure eating disorder symptoms, psychosocial impairment, self-criticism, depression and anxiety. The intervention is a 10 to 12-week closed therapy group for students seeking support regarding issues related to eating, weight and shape concerns. Group members will be facilitated to recognise and explore some of the difficult emotions underlying these issues. In particular, the group will focus on 'taming' the inner critic, that part of ourselves that criticises or chastises us for not being good enough. By identifying the critic in ourselves and by witnessing it in others, group members may be better positioned to figure out what they really need from themselves at times of difficulty. There will be some information provided around eating and emotions, with the focus of the sessions being on experiential exercises under the guidance of the group facilitators.

What are the possible disadvantages and risks of taking part? Participation in this study will involve reflecting on and talking about difficult and sensitive topics related to your eating, weight and shape concerns and self-criticism. This can sometimes lead to emotional distress. To ensure everyone feels supported, the group therapy sessions will be facilitated by experienced therapists who are trained in handling emotional distress. If you feel overwhelmed at any point, you are encouraged to communicate with the group facilitators, who can provide support and refer you to additional resources if required. Group participants are required to be respectful of other participants' concerns and difficulties and confidentiality is of paramount importance to ensure a safe environment for sharing. If you are in the control group and feel overwhelmed, you are encouraged to speak with the Student Counselling and Wellbeing Service staff involved in your support, who will be able to respond to your concerns and refer you to additional resources if required.

What are the possible benefits of taking part? By participating in this study, you may experience improvements in your relationship with food, body image, and self-criticism. Engaging in group therapy can also provide a supportive environment where you can connect with others facing similar challenges. Although benefits cannot be guaranteed, many participants find that this type of therapy helps them develop healthier coping strategies and a more compassionate view of themselves. We cannot promise the study will help you but the information we get from this study will help improve the treatment of people with eating disorders and eating, weight and shape concerns.

What if there is a problem? Any complaint about the way you have been dealt with during the study or any possible harm you might suffer will be addressed. The detailed information about this is given in Part 2 of this information sheet.

Will information from or about me from taking part in the study be kept confidential? Yes. We will follow ethical and legal practice and all information about you will be handled in confidence. There are some rare situations in which information would have to be shared with others. Details about this are included in Part 2 of this information sheet.

Part 2

What will happen if I don't want to carry on with the study? There are two possible ways of withdrawing from this study. Firstly, if you are in the intervention group, you may choose to withdraw from the group emotion-focused therapy sessions but remain willing to complete questionnaires. Secondly, participants from either group (intervention or treatment as usual control) may wish to withdraw from the study altogether. Either of these can be done at any point throughout the study without reason. If you decide to fully withdraw from the study, we will retain data up to the point of withdrawal because in RCTs it is important to have information on all participants regardless of how long they remain in the study.

What if there is a problem? If you have a concern about any aspect of this study and this has not been resolved by speaking to the group facilitators or Student Counselling and Wellbeing Service staff involved in your support in the first instance, or if it feels more appropriate to speak with the research team, the research team will do their best to address your concerns. If you remain unhappy and wish to make a formal complaint, you can do so by contacting Dr. Fergal Jones, Research Director at the Salomons Institute for Applied Psychology (contact details provided in the next section).

Concerns and Complaints If you have a concern about any aspect of this study, you can email me, as the lead researcher, and I will do their best to address your concerns. My email address is aa1428@canterbury.ac.uk If you remain unhappy and wish to complain formally, you can do this by contacting Dr Fergal Jones, Research Director, Salomons Institute for Applied Psychology: fergal.jones@canterbury.ac.uk or by leaving a message on the 24-hour voicemail phone number 01227 927070.

Will information from me or about me from taking part in this study be kept confidential? Your confidentiality is important and therefore all information collected as part of the project will be kept strictly confidential, except in the event where information is shared that suggests a risk of harm to yourself or others (in which case we would need to disclose information to a third party but would endeavour to speak with you about this first). Data collected will include your name, contact details, some demographic characteristics and answers to online questionnaires measuring eating disorder symptoms, the impact of these on your psychosocial functioning, self-criticism, depression, anxiety and stress, along with your thoughts about the helpfulness, accessibility and acceptability of the intervention if you are in the intervention group. Data will be anonymised and stored securely in accordance with data protection regulations. The lead researcher and lead supervisor will be the only people who has access to any personally identifiable information. Once we have finished the study, we will keep the data securely for ten years and then securely destroy it. You have the right to check the accuracy of data held about you and correct any errors.

What will happen to the results of the research study? Results will be included in an anonymised written report that I will submit to the Doctorate in Clinical Psychology programme at the Salomons Institute for Applied Psychology. There is the possibility that anonymised quotations from open-ended questions on questionnaires will be used in this report. There is also the possibility that the report may be published in an academic journal. If you wish to be sent a copy of the final report then you are able to request this by emailing the leader researcher (Ali Argo): aa1428@canterbury.ac.uk

Who is organising and funding the research? This study was organised by the lead researcher (Ali Argo) with input from a lead supervisor (Dr Anna Oldershaw) and secondary supervisor (Dr Daragh Keogh), as part of the lead researcher's Clinical Psychology doctoral training at Canterbury Christ Church University. Canterbury Christ Church University has funded this study.

Who has reviewed the study? All research is looked at by an independent group of people called a Research Ethics Committee, to protect your interests. This study has been reviewed and approved by the Salomons Ethics Panel, Salomons Institute for Applied Psychology, Canterbury Christ Church University.

Further information and contact details Should you require further information regarding this research project, please do not hesitate to contact me via email at aa1428@canterbury.ac.uk If you would like to speak to my lead supervisor for this study, please contact anna.oldershaw@canterbury.ac.uk

ELIGIBILITY:
Inclusion Criteria:

* 1. Open referral with the counselling/student support service, meaning students can engage in a screening appointment with a group facilitator 2. Global EDE-Q Score ≥ 2.77 (cutoff for disordered eating in the general population as per EDE-Q norms attached).

or Score ≥ Mean + 1 SD on at least one EDE-Q subscale (Restraint, Eating Concern, Shape Concern, or Weight Concern) 3. Have body mass index (BMI) greater than 15kg/m2 4. Have sufficient English for talking therapy 5. Over the age of 18

Exclusion Criteria:

* 1. Considerable psychological risk, including active suicidal plans 2. Comorbidity taking priority 3. Alcohol/substance use disorder 4. Psychosis 5. Risk of harm towards others 6. Participating in concurrent psychological one-to-one or group treatment 7. Diagnosed intellectual disability impeding ability to access therapy 8. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The Eating Disorder Examination Questionnaire (EDE-Q) | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  A 28-item self-report questionnaire, measuring the range, frequency and severity of behaviours associated with a diagnosis of an ED. It is categorised into 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and an overall global score, with a higher score indicating more problematic eating difficulties. To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscale. To obtain an overall or 'global' score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e. four). Subscale scores are reported as means and standard deviations. Likert scale ranges from 0 to 6, therefore minimum score is 0 and maximum score is 6.

SECONDARY OUTCOMES:
The Clinical Impairment Assessment Questionnaire (CIA) | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  A 26-item self-report questionnaire, measuring the severity of psychosocial impairment as the result of ED features. It is designed to be completed straight after a measure of current ED symptoms that covers the same time frame of 28 days (such as the EDE-Q). It covers impairment in domains typically affected by EDs: mood and self-perception, cognitive functioning, interpersonal functioning and work performance. Scores range from 0 to 48, with higher ratings indicate a higher level of impairment.
The Forms of Self-Criticism/Attacking & Self-Reassuring Scale (FSCRS) | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  A 22-item self-report questionnaire, measuring ways in which people think about feel about themselves when things go wrong for them. There are three factors: inadequate self, hated self and reassured self. Each item is rated on a scale from 0 to 4. Items are grouped by subscales: inadequate self, hated self, and reassured self. Higher scores on the first two of these indicate stronger self-critical or self-attacking tendencies. Higher scores on reassured self indicate better ability to self-reassure and be compassionate towards oneself. Each subscale is scored independently and there is no single combined overall score.
Depression Anxiety Stress Scales-Short Form (DASS-21) | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  A 21-item self-report questionnaire, assessing the severity of general psychological distress and symptoms related to depression, anxiety and stress. Scores are presented as a total score (between 0 and 63) and a score for the three subscales (between 0 and 21). Higher scores indicate higher levels of anxiety, depression and stress.
Counseling Center Assessment of Psychological Symptoms (CCAPS) 34 | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  The CCAPS-34 was released in September, 2009 and updated in 2012. It is a 34-item instrument with seven distinct subscales that are related to psychological symptoms and distress in college students. Higher scores represent greater distress or severity of symptoms in the specific subscale area. Scores range between 0 and 4 on each of the items.
Difficulties in Emotion Regulation Scale (DERS) | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  The Difficulties in Emotion Regulation Scale (DERS) is an instrument measuring emotion regulation problems. Scores are presented as a total score as well as a score for each of the 6 subscales. Higher scores suggest greater problems with emotion regulation. Maximum possible score 180 and minimum possible 16.
Bespoke questionnaire to measure the acceptability of the intervention | From baseline prior to the intervention/control condition beginning to post-intervention (2-4 weeks post-intervention)
  Bespoke questionnaire using Likert scales, open text responses for more information about choices given, and yes/no to recommending the intervention to other students experiencing difficulties related to an eating disorder or eating, weight and shape concerns.

CONTACTS AND LOCATIONS:
Locations (1):
- Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For participants who opt to take part in a qualitative study conducted by a fellow doctoral student, I will pass on their email addresses to this student/researcher once they have given consent.